CLINICAL TRIAL: NCT03689140
Title: Mobile Health Intervention for Family Smoking Cessation in Romania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Babes-Bolyai University (Other); University of Michigan (Other); Wake Forest University Health Sciences (Other)
Responsible Party: Principal Investigator, Cristian Meghea, Assistant Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R21TW010896 (NIH)
Record Dates: First submitted 2018-09-19; First posted 2018-09-28 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Telemedicine: Smoking Cessation App Only; Telemedicine: Smoking Cessation Counseling; Telemedicine: App + Counseling; Usual Care
Keywords: mHealth; Mobile health; Telehealth; Pregnancy; Tobacco; Cessation
MeSH Terms: interventions — Telemedicine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- App-only (Experimental): The intervention will consist of participants will only use a smoking cessation app
  Interventions: Behavioral: Smoke Free Together - App-only
- Telemedicine counseling only (Experimental): The intervention will consist of participants will only use telemedicine counseling
  Interventions: Behavioral: Smoke Free Together - Telemedicine counseling only
- App + telemedicine counseling (Experimental): The intervention will consist of participants will only use a smoking cessation app + telemedicine counseling
  Interventions: Behavioral: Smoke Free Together - app + telemedicine
- Usual Care (No Intervention): The participants will continue with usual care

INTERVENTIONS:
Behavioral: Smoke Free Together - App-only — Pregnant smokers and their life partners will use a smoking cessation app.
  Arms: App-only
Behavioral: Smoke Free Together - Telemedicine counseling only — Pregnant smokers and their life partners will use telemedicine, real time video counseling on smoking cessation
  Arms: Telemedicine counseling only
Behavioral: Smoke Free Together - app + telemedicine — Pregnant smokers and their life partners will use telemedicine and an app for smoking cessation
  Arms: App + telemedicine counseling

SUMMARY:
The objectives of this study are to determine in a randomized controlled trial (RCT) whether a mobile health (mHealth) couples intervention shows promise in increasing smoking cessation among pregnant couples who smoke and to build mHealth research capacity in Romania. The intervention will be novel in its use of the unique functionality of smartphones, its emphasis on the dyadic efficacy for smoking cessation, and the focus on pregnant couples. Our aims are to (1) Test the implementation feasibility, acceptability, and initial efficacy of a culturally-adapted mHealth smoking cessation intervention among couples during pregnancy and postpartum in Romania. (2) Develop mHealth research capacity by enhancing individual and institutional research capabilities in Romania and expanding the existing international research network.

ELIGIBILITY:
Inclusion Criteria:

* pregnant smokers in the 2nd or 3rd pregnancy trimester and their partners.
* 18 years or older
* married or in a stable relationship
* owns and uses an Android smartphone with broadband internet connection
* willing to have the partner contacted for participation.

Exclusion Criteria:

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 324 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2020-08-24 (Actual); Study Completion 2020-08-24 (Actual)

PRIMARY OUTCOMES:
Percentage of women in each arm who stopped smoking, and who relapsed smoking postpartum | Change from smoking at baseline to quitting assessed at 3 months after the intervention is completed
  The primary outcomes are maternal pregnancy smoking cessation and postnatal relapse. Maternal smoking status will be biochemically verified at the final follow-up based on salivary cotinine obtained by mail.

CONTACTS AND LOCATIONS:
Locations (1):
- Babes-Bolyai University, Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Informed Consent Form: Informed consent for women (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/40/NCT03689140/ICF_000.pdf
  • Informed Consent Form: Informed consent for partners (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/40/NCT03689140/ICF_001.pdf